CLINICAL TRIAL: NCT00429221
Title: ADHD Medication Adherence: A Parent-Provider Intervention Modeled From HIV
Brief Title: Parent-Provider Intervention for Improving Medication Adherence in Children With Attention Deficit Hyperactivity Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: #5327; R34MH078700 (NIH); DAHBR 96-BHA
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

INTERVENTIONS:
Behavioral: Tailored Medication Messages for Parents

SUMMARY:
This three-phase study will develop and test a provider-administered intervention to improve medication adherence and promote sustained medication use among children with ADHD and their caregivers.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is a common childhood behavior disorder that causes impaired functioning in multiple settings, including home, school, and in relationships with peers. Symptoms of ADHD include impulsiveness, hyperactivity, and inattention. Both medications and behavior therapies have been shown to be effective in treating ADHD. It is essential, however, that children take their medication regularly for it to be effective. This three-phase study will develop and test a provider-administered intervention to improve medication adherence and persistence among children with ADHD and their caregivers.

The first phase of this study will gather information about perspectives on ADHD and its treatment by using focus groups and interviews with participating children and their parents. Phase two of the study will gather information on medication adherence and persistence, as well as demographic information. Phase three of the study will involve developing and testing a three part intervention consisting of an ADHD education component, a short survey to help parents identify non-adherence warning signs, and tailored medication messages for parents. After conducting a pilot with five parent-child pairs to assess feasibility and accessibility, all interested doctors at the study site will receive a lecture on evidence-based treatments for ADHD and a supply of parent ADHD education toolkits. Half of the doctors will be randomly assigned to receive additional training on the experimental procedures and to administer the intervention as part of the study. Parent and child participants will be randomly assigned to receive either treatment with a doctor who has been trained on the experimental intervention or treatment as usual. Assessments will take place at the beginning of treatment and 1, 3, and 6 months after the start of treatment. During each assessment, a saliva sample will be collected from the child, and parents will complete several checklists and questionnaires about ADHD treatment and medication adherence.

ELIGIBILITY:
PHASE I:

Inclusion Criteria:

Parent Focus Group Participants:

* Must be primary caregiver and legal guardian of child (6-10 years) at time of initial ADHD diagnosis
* Child must have been diagnosed with ADHD within the last 18 months at Schneider Children's Hospital's (SCH) outpatient clinic (co-morbid diagnosis of oppositional defiant disorder [ODD] or conduct disorder [CD] is permitted)

Provider Focus Group Participants:

* Child psychiatrist employed by North Shore - Long Island Jewish child psychiatry outpatient department
* Licensed to practice in New York State
* Has more than 1 year of experience prescribing medication to youth with ADHD

Child Interview Participants:

* Diagnosis of ADHD (co-morbid diagnosis of ODD, CD, or mood disorder is permitted)
* Between 6 and 10 years old at time of initial ADHD diagnosis
* Diagnosis occurred within 18 months prior to study entry at Zucker Hillside Hospital outpatient clinic

Exclusion Criteria:

Parent Focus Group Participants and Child Interview Participants:

* Child has significant co-morbid medical conditions, such as diabetes, cystic fibrosis, or severe asthma, resulting in more than 2 emergency visits in the last year
* Child has a co-morbid diagnosis of psychosis, bipolar disorder, or other serious psychiatric condition within 12 months prior to study entry
* Child has history of psychiatric hospitalization within 12 months prior to study entry
* Child is receiving treatment in a different setting

PHASE II:

Inclusion Criteria:

* Primary caregiver and legal guardian of child (6-10 years) at the time of initial ADHD diagnosis
* Child has been diagnosed with ADHD within the last 18 months at SCH's outpatient clinic

Exclusion Criteria:

* Parents of children with co-morbid medical conditions other than oppositional defiant disorder (ODD) or conduct disorder (CD)
* Parents of children with a co-morbid diagnosis of psychosis, bipolar disorder, mental retardation, or other severe mental illness, evidence of mental retardation, or history of psychiatric hospitalization within 12 months prior to study entry
* Child is receiving treatment in a different setting

PHASE III:

Inclusion Criteria:

* Medication naïve children with a primary diagnosis of ADHD (co-morbid ODD will be permitted) at the Child Psychiatric Outpatient Department at SCH
* Parents are the legal guardians
* Both parents and children willing to sign the informed consent/assent

Exclusion Criteria:

* Children with co-morbid medical conditions other than ODD
* Children with a co-morbid diagnosis of psychosis, bipolar disorder, or other serious psychiatric condition, evidence of mental retardation, or history of recent hospitalization

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01

PRIMARY OUTCOMES:
Parents' attitudes and beliefs
Parents' reported adherence, prescription refill, and side effect information
Children's adherence (all measured at Months 1, 3, and 6)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Pappadopulos, PhD, Principal Investigator — Columbia University/New York State Psychiatric Institute

REFERENCES:
- [Background] Rizzo JA, Simons WR. Variations in compliance among hypertensive patients by drug class: implications for health care costs. Clin Ther. 1997 Nov-Dec;19(6):1446-57; discussion 1424-5. doi: 10.1016/s0149-2918(97)80018-5. PMID 9444452
- [Background] Dolezal C, Mellins C, Brackis-Cott E, Abrams EJ. The reliability of reports of medical adherence from children with HIV and their adult caregivers. J Pediatr Psychol. 2003 Jul-Aug;28(5):355-61. doi: 10.1093/jpepsy/jsg025. PMID 12808012
- [Background] Mellins CA, Brackis-Cott E, Dolezal C, Abrams EJ. The role of psychosocial and family factors in adherence to antiretroviral treatment in human immunodeficiency virus-infected children. Pediatr Infect Dis J. 2004 Nov;23(11):1035-41. doi: 10.1097/01.inf.0000143646.15240.ac. PMID 15545859
- [Background] Achenbach TM, Howell CT, Quay HC, Conners CK. National survey of problems and competencies among four- to sixteen-year-olds: parents' reports for normative and clinical samples. Monogr Soc Res Child Dev. 1991;56(3):1-131. PMID 1770964
- [Background] Swanson J, Nolan R, Pelham W (1988): Swanson, Nolan and Pelham rating scale (SNAP). Pittsburgh, PA, Department of Psychiatry, Western Psychiatric Institute and Clinic.
- [Background] Hollingshead, A. B. (1975). Four factor index of social status. Unpublished manuscript, Yale University, NewHa ven, CT.